CLINICAL TRIAL: NCT06474754
Title: Enhancing Precise Perioperative Risk Surveillance: Validation of Submaximal Cardiopulmonary Exercise Testing to Usual Care for Detection of Myocardial Injury After Noncardiac Surgery
Brief Title: Submaximal Cardiopulmonary Exercise Testing for Detection of Myocardial Injury After Noncardiac Surgery
Acronym: EnhanceMINS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000037991
Record Dates: First submitted 2024-06-14; First posted 2024-06-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Myocardial Injury After Non-cardiac Surgery; Submaximal Exercise Performance; Preoperative Period
Keywords: submaximal cardiopulmonary exercise testing; MINS; myocardial injury after noncardiac surgery; perioperative myocardial injury; anesthesiology

STUDY DESIGN:
Intervention Model Description: Single-blinded Phase IV diagnostic clinical trial study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Submaximal cardiopulmonary exercise testing (Experimental): Single arm design; selected participants will receive both usual care (Duke Activity Status Index) and submaximal cardiopulmonary exercise testing. All participants will receive high-sensitivity troponin measurements on operative day 1 and postoperative day 1,2,3
  Interventions: Diagnostic Test: High-sensitivity troponin, serum; Diagnostic Test: Submaximal Cardiopulmonary Exercise Testing; Diagnostic Test: Duke Activity Status Index

INTERVENTIONS:
Diagnostic Test: High-sensitivity troponin, serum — A serum derived measure of myocardial injury. Threshold value of 14ng/L.
  Other Names: HST
Diagnostic Test: Submaximal Cardiopulmonary Exercise Testing — FDA-approved device uses breath by breath sampling during calibration and exercise challenge. Analysis is performed using a differential pressure pneumotach method for volume calibration and measurement, an infrared sensor for CO2 and a paramagnetic sensor for O2 measurements. Automated calibration using a calibration gas mixture (15.6% O2/5% CO2) is performed at regular intervals. The Shape II calculations used to differentiate causes of exertional dyspnea are Artificial Intelligence (AI) based algorithms and measurements have been previously validated to conventional cardiopulmonary exercise testing methods. Brief smCPET is comprised of a 2-minute calibration phase, 3 minutes of graded exercise using a stair-step and a 1 minute recovery phase for a total of 6 minutes. An instant report is then generated.
  Other Names: smCPET
Diagnostic Test: Duke Activity Status Index — A validated measure of preoperative functional capacity which will be utilized to cross-validate smCPET peak VO2. Low DASI score has been found to estimate peak oxygen uptake (VO2), predict MINS, myocardial infarction, and inducible myocardial ischemia on myocardial perfusion scintigraphy.
  Other Names: DASI

SUMMARY:
The goal of this clinical trial is to learn whether physicians can associate evidence of myocardial injury after surgery with findings obtained from submaximal cardiopulmonary exercise testing. The main questions are:

Is detection of postoperative myocardial injury with submaximal cardiopulmonary exercise testing superior to using usual care?

And which submaximal cardiopulmonary exercise testing measure is better?

Participants will undergo evaluation with a short submaximal cardiopulmonary exercise test, then undergo surgery. Myocardial injury will be measured on postoperative days 0, 1, 2, and 3 (during and up to 3 days after surgery). These results will analyzed by comparing it to findings from the submaximal cardiopulmonary exercise test.

If there is a relationship, this will help anesthesiologists and surgeons assign certain treatments that may reduce the risk of developing myocardial injury after surgery.

DETAILED DESCRIPTION:
Among the 50 million US adults undergo non-cardiac surgery each year, an estimated 1.4-3.9% of patients experience perioperative myocardial infarction with another 6-18% showing evidence of myocardial injury. These cardiac insults, known as myocardial injury after noncardiac surgery (MINS) are associated with a 2.7-3.2 fold higher odds of 30-day mortality, 2.2 fold higher odds of nonfatal myocardial infarction (MI), 1.55 fold increase in 30-day congestive heart failure events, and 5.2 times higher risk of stroke, highlighting the importance of predicting and treating their occurrence. MINS is treatable, and potentially preventable, by a combination of tailored intraoperative monitoring and appropriate post-operative care.

The current approach to preoperative risk stratification is predominately derived from patient-reported functional capacity associated with history, physical examination and select laboratory investigations. This approach results in significant healthcare worker time and cost expenditures, without improved perioperative outcomes. In contrast, a technological approach utilizing conventional cardiopulmonary exercise testing (CPET) has been shown to improve individualized identification of high-risk patients prior to surgery. Widespread cardiopulmonary exercise test adoption in the perioperative setting, however, has been limited by cost, technical requirements, and time investment despite its documented utility in cardiopulmonary risk assessment. However, brief submaximal cardiopulmonary exercise testing (smCPET) addresses the limitations of conventional CPET including low cost, low time investment, small footprint, and ease of operator efficiency. In our pilot (under review), we demonstrated the feasibility and performance of implementing smCPET within a high-volume pre-surgical evaluation clinic.

This proposal seeks to continue work in characterizing smCPET and its role in individualized preoperative risk identification. The aim of this study proposal is to validate two clinically relevant questions: 1) Are smCPET measures superior to usual care (Duke Activity Status Index) in patients undergoing moderate to high-risk noncardiac surgery and 2) to determine which smCPET measure is more sensitive to MINS as described by abnormalities in postoperative high-sensitivity troponin measurements.

Using a smCPET-guided approach, this study seeks to characterize its value in identifying high-risk patients for MINS, provide further validation of smCPET utility as a preoperative risk stratification approach, and preliminarily identify smCPET measures with highest association with MINS.

If validated, this would provide the foundation for a smCPET-guided clinical decision support system of preoperative identification and perioperative monitoring that could 1) enhance patient outcomes by providing early prediction and detection of MINS and 2) characterize a research methodology to stratify participants for further research in assessing perioperative strategies to reduce MINS. These findings will provide one of the first examples of quantitative and individualized preoperative risk identification methods for a common and deleterious perioperative outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Biological male or female, aged 45 years or older.
4. In good general health as evidenced by medical history or diagnosed with metabolic equivalents (self-reported ability to climb 1 flight of stairs).
5. Revised Cardiac Risk Index less than or equal to three.
6. Willing to accept phlebotomy on operative day 0, 1, 2, and 3, as part of usual care.
7. Scheduled for moderate to high-risk elective non-cardiac surgery with an expected 24-72 hour stay within 60 days of enrollment in the study.

Exclusion Criteria:

1. Inability to perform study procedures as defined by inability to achieve greater than 4 metabolic equivalents (cannot climb 1 flight of stairs reliably).
2. Pregnancy or lactation.
3. Inability to give independent informed consent.
4. Revised cardiac risk index greater than 3.
5. Recent myocardial infarction (less than 6 weeks).
6. Recent anginal symptoms (stable or unstable) within past 6 months.
7. Recent admission or endorsement for congestive heart failure within 6 months
8. Recent admission or endorsement for syncope within 6 months.
9. Symptomatic tachy- or bradyarrhythmia (supraventricular tachcardia, ventricular tachycardia with symptoms of intermittent dizziness, pre- syncopal events)
10. Uncorrected severe valvular heart disease (severe aortic, tricuspid or mitral stenosis)
11. Acute pulmonary embolism or deep vein thrombosis (within past 6 months)
12. Uncontrolled pulmonary edema
13. Uncontrolled symptomatic cardiac arrhythmias.
14. Active endocarditis
15. Active myocarditis or pericarditis
16. Active wheezing or recent exacerbation of chronic obstructive pulmonary disease admission in past 6 months.
17. Inability to perform components of the SHAPE test (severe hip flexion limitation, severe osteoarthritis of knee or hip, limb immobilization, ambulation requires cane or crutches, baseline balance irregularities.
18. Diagnosis of symptomatic vertigo
19. Known allergic reactions to components of the SHAPE medical system apparatus disposable mouthpiece.
20. Active enrollment in an interventional clinical trial within the enrollment period of the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
MINS | Operative Day 0, Postoperative Day 1, 2 or 3
  Myocardial Injury after noncardiac surgery. Measurement: High-Sensitivity Troponin assay with an abnormal value defined as 14 nanograms per liter or greater.

SECONDARY OUTCOMES:
30-day Major Adverse Cardiovascular Events | Postoperative Day 1 through Postoperative Day 30
  30-day recorded events of atrial fibrillation, angina, stroke, myocardial infarction, congestive heart failure as defined by International Classification of Disease (Version 10) coding.
Length of Stay | From operative day 0 through hospital discharge up to postoperative day 180
  Measurement of patient inpatient status from operative day 0 through physical discharge from the hospital.
Readmission | Postoperative Day One through Postoperative Day 60.
  Readmission of any type from the time of surgical procedure discharge through postoperative day 60.

CONTACTS AND LOCATIONS:
Overall Officials: Zyad J Carr, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University; Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, informed consent and human study record will be provided. A deidentified dataset will be uploaded to the data sharing repository NIBIB physionet website.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: For 24 months after initial study publication.
Access Criteria: CITI trained certified individuals that meet criteria set forth by physionet.org.
URL: https://www.physionet.org

REFERENCES:
- [Background] Snowden CP, Prentis JM, Anderson HL, Roberts DR, Randles D, Renton M, Manas DM. Submaximal cardiopulmonary exercise testing predicts complications and hospital length of stay in patients undergoing major elective surgery. Ann Surg. 2010 Mar;251(3):535-41. doi: 10.1097/SLA.0b013e3181cf811d. PMID 20134313
- [Background] Le Manach Y, Perel A, Coriat P, Godet G, Bertrand M, Riou B. Early and delayed myocardial infarction after abdominal aortic surgery. Anesthesiology. 2005 May;102(5):885-91. doi: 10.1097/00000542-200505000-00004. PMID 15851872
- [Background] Devereaux PJ, Goldman L, Cook DJ, Gilbert K, Leslie K, Guyatt GH. Perioperative cardiac events in patients undergoing noncardiac surgery: a review of the magnitude of the problem, the pathophysiology of the events and methods to estimate and communicate risk. CMAJ. 2005 Sep 13;173(6):627-34. doi: 10.1503/cmaj.050011. PMID 16157727
- [Background] Patel AY, Eagle KA, Vaishnava P. Cardiac risk of noncardiac surgery. J Am Coll Cardiol. 2015 Nov 10;66(19):2140-2148. doi: 10.1016/j.jacc.2015.09.026. PMID 26541926